# Title: Effects of High Amplitude and Focused tACS on Entraining Physiological Tremor

Date: 01-June-2016

## Protocol unfocused electrodes - Healthy volunteers

- 1. Patient consent (20 min)
  - a. Explain the study
  - b. Let subject read & fill in informed consent
- 2. Patient preparation (1h)
  - a. Clean big regions of the scalp with ethanol around the left motor cortex and the prefrontal cortex
  - b. Measure Cz, C1 and C3 and place the stimulating electrode between C1 and C3.
  - c. Place another stimulating electrode over the PFC (by measuring F5/F6)
  - d. Place the return electrode over the ankle
  - e. Calibrate the accelerometer
  - f. Place the accelerometer on the middle finger of dominant hand
  - g. Ask subject to adopt a tremor inducing pose
  - h. Measure the tremor frequency for 5 minutes and analyse with specTremor
  - i. Check if impedance is below  $5k\Omega$
  - j. If impedance is too high, add more saline
- 3. Stimulation amplitude dose response (10 min)
  - a. Instruct the subject to report any stimulation related side effects / secondary effects (tingling, pain, phosphenes)
  - b. Apply stimulation with increasing currents, while
    - i. Monitoring impedance
    - ii. Asking the subject about side effects
  - c. As long as no severe side effects are reported and subject wants to increase the current, increase with small steps (e.g. 0.2 mA) until a maximum of 2mA.
  - d. Repeat for second stimulation site
  - e. Determine the maximal amplitude that is tolerable in both regions. So stimulate the two regions at the same amplitude.
- 4. Phosphene ratings and thresholds (10 min)
  - a. Check phosphene ratings at maximal stimulation amplitude for both stimulation sites
  - b. If phosphenes are reported, determine the phosphene thresholds for both sites by gradually increasing the stimulation amplitude
- 5. Stimulation protocol (45 min)
  - a. Measure the tremor frequency
  - b. Perform the stimulation protocol at the maximum stimulation amplitude determined in step 3.
  - c. Record one session of 30 sec OFF-1 min MC-30 sec OFF-1 min PFC repeated 4 times in random order
  - d. Repeat 2 more times to have 3 sessions

## **Protocol focused electrodes - Healthy volunteers**

- 6. Patient consent (20 min)
  - a. Explain the study
  - b. Let subject read & fill in informed consent
- 7. Patient preparation (1h)
  - a. Clean big regions of the scalp with ethanol around the left motor cortex and the occipital cortex
  - b. Place the electrode cap over the head of the subject
  - c. Measure if Cz of the cap matches the position of the vertex
  - d. Indicate with marker the position of the stimulating electrodes
  - e. Remove the electrode cap
  - f. Measure if the stimulating electrode is at the correct position (C3). If not, repeat a-e.
  - g. Apply EMLA-cream around the stimulating electrode positions
  - h. Calibrate the accelerometer
  - i. Place the accelerometer on the middle finger of dominant hand
  - j. Ask subject to adopt a tremor inducing pose
  - k. Measure the tremor frequency for 5 minutes and analyse with specTremor
  - I. After half an hour after applying the EMLA cream, check if the hair is dry. If the hair is still too wet, dry with paper/towel or a hairdryer.
  - m. Place the electrode cap over the head of the subject
  - n. Measure the head to ensure that the location of the motor cortex matches the position of the plastic electrode holders.
  - o. Add electrolyte gel inside the electrode holders with a syringe
    - i. 2.5 ml for flat electrode holders
    - ii. 5 ml for Gamma
  - p. Add the electrodes and close the electrode holders
  - q. Check if impedance is below  $5k\Omega$
  - r. If impedance is too high, add more gel or attach rubber straps over the electrodes for good contact of the electrode holders and the scalp.
- 8. Stimulation amplitude dose response (10 min)
  - a. Instruct the subject to report any stimulation related side effects / secondary effects (tingling, pain, phosphenes)
  - b. Apply stimulation with increasing currents, while
    - i. Monitoring impedance
    - ii. Asking the subject about side effects

- c. As long as no severe side effects are reported and subject wants to increase the current, increase with small steps (e.g. 0.5 mA) until a maximum of 5mA.
- d. Repeat for second stimulation site
- e. Determine the maximal amplitude that is tolerable in both regions. So stimulate the two regions at the same amplitude.
- 9. Phosphene ratings and thresholds (10 min)
  - a. Check phosphene ratings at maximal stimulation amplitude for both stimulation sites
  - b. If phosphenes are reported, determine the phosphene thresholds for both sites by gradually increasing the stimulation amplitude

### 10. Stimulation protocol (45 min)

- a. Measure the tremor frequency
- b. Perform the stimulation protocol at the maximum stimulation amplitude determined in step 3.
- c. Record one session of 1min OFF-1 min MC-1 min OFF-1 min OC repeated 3 times in random order
- d. Repeat 2 more times to have 3 sessions

#### **Statistics**

Statistics are performed with a significance level  $\alpha$ =0.05. A two-sided Wilcoxon signed-rank test compares scores for phosphene intensity and thresholds between the different conditions. For phase entrainment the effect of the condition on the entrainment is tested with a non-parametric Friedman test. If significant, a post-hoc analysis is conducted with a two-sided Wilcoxon Signed-Rank test between all pairs of the conditions. p-values are adjusted for multiple comparisons with a Bonferroni correction.